CLINICAL TRIAL: NCT05524935
Title: A Phase II Trial of Olaparib in Combination With Pembrolizumab for Advanced Uveal Melanoma
Brief Title: Olaparib in Combination With Pembrolizumab for Advanced Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21731; 58050 (Other: Merck & Co, Inc.)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma; Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab and Olaparib (Experimental): Participants will be given 200 mg Pembrolizumab IV every 21 days + will take 300 mg Olaparib by mouth twice daily days 1-21 of each 21 day cycle. Treatment will continue until progression, unacceptable toxicity, or for a maximum of 35 treatment cycles
  Interventions: Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab Day 1 of each 21 day (3 week) cycle
  Other Names: Keytruda
Drug: Olaparib — Olaparib by mouth days 1-21 of each 21 day (3 week) cycle
  Other Names: AZD2281; KU-0059736; Lynparza

SUMMARY:
This is a prospective phase II multi-center trial of the combination of the PARP inhibitor olaparib with the immune checkpoint inhibitor pembrolizumab in advanced uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic uveal melanoma will be enrolled in this study. Prior hepatic directed therapy for metastatic uveal melanoma is permitted.
* Male participants: A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 200 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies: (a) Not a woman of childbearing potential (WOCBP) as defined in Appendix 3, OR (b) A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1.49 Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have the ability to swallow oral medications (olaparib).
* Have adequate organ function as defined in the protocol.

Exclusion Criteria:

* A woman of childbearing potential (WOCBP) who has a positive urine or serum pregnancy test within 72 hours prior to start of study therapy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent as monotherapy or as combination therapy for uveal melanoma. Note: these agents may have been used for the treatment of another malignancy as long as the therapy was completed more than 2 years ago (calculated from the date of signing the ICF).
* Has received prior PARP inhibitor therapy.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [or 5 half-lives of the agent, whichever is shorter] prior to planned start of study therapy. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline (with the exception of endocrine toxicity requiring replacement therapy which is permissible)
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent; for CNS metastases, see permissible steroid dosing in exclusion criterion #9 below) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or requires active treatment, the lack of which would pose a risk to the health of the subject, in the opinion of the investigator.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and using no more than the equivalent of 2mg daily of dexamethasone (or equivalent corticosteroid).
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: this is by history; testing is not required unless clinically suspected
* Has a known history of active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: testing for Hepatitis B and Hepatitis C is not required unless clinically indicated or mandated by local health authority.
* Has a known history of active tuberculosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 24 months
  Overall Response Rate is defined as the rate of the best overall response as complete response (CR) +partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months
  Progression Free Survival is defined as the time from start of treatment to first documentation of disease progression, death, or change of treatment. Participants receiving ongoing therapy at the time of data analysis will be censored.
Overall Survival (OS) | up to 24 months
  Overall survival will be calculated from the start of treatment until death from any cause. Participants alive at the time of data analysis will be censored.
Number of Adverse Events related to study treatment | up to 24 months
  All toxicity analyses will be collated according to grade and frequency. This will include all events considered possibly, probably, or definitely related to study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil I Khushalani, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided